CLINICAL TRIAL: NCT02775656
Title: An Observational Follow-up Study of Women Who Become Pregnant While Participating in a Certolizumab Pegol (CZP) Clinical Study or Whose Pregnancies Have Otherwise Been Reported to UCB Due to Potential CZP Exposure During Pregnancy
Brief Title: UCB Cimzia Pregnancy Follow-up Study
Status: Terminated | Type: Observational
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Collaborators: Syneos Health (Other); Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: UP0019
Record Dates: First submitted 2016-03-08; First posted 2016-05-17 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Rheumatoid Arthritis (RA); Crohn's Disease (CD); Psoriatic Arthritis (PsA); Axial Spondyloarthritis and Ankylosing Spondylitis
Keywords: Cimzia®; CZP; Pregnancy Follow up study; Autoimmune diseases; Pregnancy outcomes; major congenital malformations; birth outcomes; malformation; birth defect
MeSH Terms: conditions — Arthritis, Rheumatoid; Crohn Disease; Arthritis, Psoriatic; Axial Spondyloarthritis; Spondylitis, Ankylosing; Autoimmune Diseases; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prospective cohort: For a pregnancy to be enrolled in the prospective cohort, the pregnancy outcome cannot be known (ie, no prenatal diagnosis of a fetus with a congenital defect and the pregnancy is still ongoing at the time of consent).
- Retrospective cohort: For a pregnancy to be enrolled in the retrospective cohort, the pregnancy outcome must already be known (ie, a congenital defect has already been identified at the time of consent into the pregnancy follow-up study, or the pregnancy has been completed at the time of consent).

SUMMARY:
The purpose of this observational follow-up study is to collect data systematically on pregnancies and offspring of women who become pregnant while participating in a Certolizumab Pegol (CZP) study or whose pregnancies have otherwise been reported to UCB due to potential CZP exposure during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy is identified while the patient is participating in an interventional or noninterventional Certolizumab Pegol (CZP) study conducted by UCB, or a development partner, regardless of phase or treatment arm (ie, commercial or investigational, placebo or comparator treatment), or whose pregnancies were spontaneously reported to UCB due to potential CZP exposure during pregnancy
* Sufficient information to classify the pregnancy as prospective or retrospective is available
* Full initial reporter (ie, woman or healthcare provider (HCP)) contact information reported to allow for follow-up (name, address, telephone number/email address) and contact information for at least 1 applicable HCP if initial contact is the woman
* Consent to participate is provided

Exclusion Criteria:

* Pregnancies in which the resulting infant is over 1 year of age at the time of informed consent will not be eligible to participate in the study

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of women who become pregnant while enrolled in a Certolizumab Pegol (CZP) study, or whose pregnancies otherwise are reported to UCB due to potential CZP exposure during pregnancy, and any resulting offspring. All pregnancies reported while the patient is enrolled in the CZP study are eligible regardless of treatment arm in the CZP study (eg, commercial or investigational CZP, placebo, or comparator treatment), pregnancy outcome (eg, live birth,spontaneous abortion, induced abortion, stillbirth) or any treatment decisions following discontinuation from the clinical study or report of the pregnancy.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Percentage of newborns with major congenital malformations | At 20 weeks gestation or greater
  The prevalence of major congenital malformations (MCMs) reported will be calculated by dividing the number of offspring with MCMs by the total number of live births and fetal losses with an MCM for all enrolled pregnancies and then stratified by treatment during pregnancy. The prevalence of MCMs will be calculated as soon as there are at least 50 prospectively-enrolled patients with an available outcome. Stillbirths and induced abortions (at 20 weeks gestation or greater) with reported MCMs are included in the estimate of the MCM prevalence.
Percentage of pregnancy outcomes with major congenital malformations | Estimated date of delivery (EDD) up to 6 weeks post-EDD
  The pregnancy outcomes with and without MCMs will be summarized using frequency counts by all trimesters of exposure and earliest trimester of exposure.

SECONDARY OUTCOMES:
Numbers of maternal pregnancy-related events | During pregnancy up to Week 40
  Descriptive statistics will be presented for the numbers of maternal pregnancy-related adverse events (AEs), adverse birth. Frequencies and proportions of adverse pregnancy will be presented using descriptive statistics. Analyses may include (but are not limited to) stratification by trimester of exposure, gestational age at time of consent, maternal age, and geographic region.
Percentage of Vaginal and C-section deliveries | At birth (Day 0)
Gestational age at birth | Estimated date of delivery (EDD) up to 6 weeks post-EDD
Birth weight | Estimated date of delivery (EDD) up to 6 weeks post-EDD
Small for gestation age | Estimated date of delivery (EDD) up to 6 weeks post-EDD
Percentage of adverse events in infants | Within the first 18 months of life
  Percentage of adverse events (AEs) being collected in infants at study follow-up period (first 18 months)
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to weight (based on the relevant population norm for the infant) | At birth (Day 0)
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to height (based on the relevant population norm for the infant) | At birth (Day 0)
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to head circumference (based on the relevant population norm for the infant) | At birth (Day 0)
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to weight (based on the relevant population norm for the infant) | 4 months
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to height (based on the relevant population norm for the infant) | 4 months
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to head circumference (based on the relevant population norm for the infant) | 4 months
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to weight (based on the relevant population norm for the infant) | 12 months
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to height (based on the relevant population norm for the infant) | 12 months
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to weight (based on the relevant population norm for the infant) | 18 months
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to height (based on the relevant population norm for the infant) | 18 months
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to gross motor skills | At birth (Day 0)
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to gross motor skills | 4 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to gross motor skills | 12 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to gross motor skills | 18 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to fine motor skills | At birth (Day 0)
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to fine motor skills | 4 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to fine motor skills | 12 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to fine motor skills | 18 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to language | At birth (Day 0)
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to language | 4 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to language | 12 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to language | 18 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to cognitive skills | At birth (Day 0)
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to cognitive skills | 4 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to cognitive skills | 12 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to cognitive skills | 18 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to social skills | At birth (Day 0)
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to social skills | 4 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to social skills | 12 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.
Percentage of infants less than or equal to the 10th percentile for sex and age with respective to social skills | 18 months
  Assessment of developmental milestones is carried out based on patient or physician report of development milestones met (Yes/No answer). 'Yes' indicates 'milestone met'; 'No' indicates 'milestone not met'.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB Pharma
Locations (1):
- Up0019 001, Wilmington, North Carolina, United States

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm